CLINICAL TRIAL: NCT04564521
Title: The Effect of Nitroglycerin on the Incidence of Cardiorespiratory Side Effect During the Intra-arterial Chemotherapy in Pediatric Patients With Retinoblastoma: a Randomized, Double-blind, Placebo-controlled, Crossover Study
Brief Title: Nitroglycerin for Intra-arterial Chemotherapy in Pediatric Retinoblastoma.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-108-1134
Record Dates: First submitted 2020-09-02; First posted 2020-09-25 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Retinoblastoma
Keywords: Intra-arterial chemotherapy; Cardio-respiratory side effects; Nitroglycerin
MeSH Terms: conditions — Retinoblastoma | interventions — Nitroglycerin; Saline Solution

STUDY DESIGN:
Intervention Model Description: Prior to the procedure, each patient will be randomized into either the saline-first arm or nitroglycerin-first arm.
  At the first intra-arterial chemotherapy after enrollment, saline or nitroglycerin is used according to the group allocation.
  At the second intra-arterial chemotherapy after enrollment, nitroglycerin is used for the saline-first arm, and saline is used for the nitroglycerin-first arm.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitroglycerin (Experimental): Intravenous nitroglycerin (0.5mcg/kg/min) is infused after the induction of general anesthesia and during intra-arterial chemotherapy.
  Interventions: Drug: Nitroglycerin
- Normal saline (Active Comparator): Normal saline is infused after the induction of general anesthesia and during intra-arterial chemotherapy.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Nitroglycerin — Intravenous nitroglycerin (0.5mcg/kg/min) is infused after the induction of general anesthesia and during intra-arterial chemotherapy to reduce the cardio-respiratory side effects.
  Other Names: Intravenous nitroglycerin
  Arms: Nitroglycerin
Drug: Normal saline — Intravenous normal saline is infused after the induction of general anesthesia and during intra-arterial chemotherapy as an active comparator.
  Other Names: Intravenous normal saline
  Arms: Normal saline

SUMMARY:
The primary objective of the study is to evaluate the effect of intravenously infused nitroglycerin on the incidence of the cardio-respiratory side effects during the intra-arterial chemotherapy for retinoblastoma in pediatric patients.

The intra-arterial chemotherapy at the ophthalmic artery is an important treatment option for retinoblastoma. However, the cardio-respiratory side effects (sudden onset of bradycardia, hypotension, a severe decrease in the compliance of lung, hypoxia) occasionally occurs during catheter manipulation in the ophthalmic artery. One of the purported mechanisms of cardio-respiratory side effects is vagal activation from the activation of trigeminal ganglion by afferent signals from the ophthalmic artery. Additionally, the chemotherapy agent can cause intra-arterial retinal precipitates. Therefore, it is expected that the dilation of the retinal artery may reduce the cardio-respiratory side effects and intra-arterial retinal precipitates.

The hypothesis of this study is that the intravenously infused nitroglycerin will increase the compliance of the ophthalmic and retinal artery and decrease vagal stimulation and cardio-respiratory side effects during catheter manipulation and chemotherapy agent infusion. This is a single-center, double-blind, randomized, placebo-controlled study comparing the effect of intravenously infused nitroglycerin and saline on the incidence of the cardio-respiratory side effect in pediatric retinoblastoma patients undergoing intra-arterial chemotherapy. Prior to the procedure, each patient will be randomized into either the control-first arm, saline, or study-first arm, nitroglycerin.

ELIGIBILITY:
Inclusion Criteria:

* Retinoblastoma patients who need intra-arterial chemotherapy under general anesthesia
* Residual intra-arterial chemotherapy ≥ 2 times (cross-over design)

Exclusion Criteria:

* Respiratory disease causing a decrease in lung compliance
* Unstable vital sign, significant arrhythmia or hypotension, Shock
* Hypersensitivity or contraindication to nitroglycerin
* Increased intracranial pressure, Intracranial hemorrhage
* Recent use of PDE5 inhibitors (<24 hours after sildenafil or vardenafil; <48 hours after tadalafil)

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of the cardio-respiratory side effects during ophthalmic artery selection and intra-arterial injection of chemotherapy agents. (percent) | During the intra-arterial chemotherapy (up to 4 hour)
  Bradycardia (< 80% of Baseline), Hypotension (< 80% of Baseline), Decrease in the lung compliance, Abnormal end-tidal CO2 curve, or Desaturation (SpO2 <95%)

SECONDARY OUTCOMES:
The duration of the cardio-respiratory side effects during ophthalmic artery selection and intra-arterial injection of chemotherapy agents. (percent) | During and after the intra-arterial chemotherapy (up to 48 hour)
  Duration between the onset and the recovery from cardio-respiratory side effects.
The incidence of using vaso-active drugs (percent) | During and after the intra-arterial chemotherapy (up to 48 hour)
  The incidence of using vaso-active drugs (e.g. vasopressor, inotropics)(percent)
The incidence of the side effect of nitroglycerin infusion (percent) | During the intra-arterial chemotherapy (up to 4 hour)
  Hypotension (< 80% of baseline) after 10 minutes from nitroglycerin infusion, or allergic reaction, etc.
The concentration of inhaled sevoflurane (vol%) | During the intra-arterial chemotherapy (up to 4 hour)
  The concentration of inhaled sevoflurane
The depth of anesthesia | During the intra-arterial chemotherapy (up to 4 hour)
  The depth of anesthesia (bispectral index or patient sedation index, 0-100, 0 smaller score means deep anesthesia and larger score means awake state.)
Duration of anesthesia (min) | During the intra-arterial chemotherapy (up to 4 hour)
  Duration of anesthesia
Total procedure time (min) | During the intra-arterial chemotherapy (up to 4 hour)
  From ophthalmic artery selection to the end of intra-arterial injection.
The procedural satisfaction score of radiologist (1-3) | During the intra-arterial chemotherapy (up to 4 hour)
  3 grades (1:poor, 2:fair, 3:good)
Incidence of the newly developed focal ischemia or infarct in retina photography(yes or no) | After the intra-arterial chemotherapy (up to 6 month)
  Incidence of the newly developed focal ischemia or infarct in retina photography(yes or no) on ophthalmology outpatient clinic after the intra-arterial chemotherapy assessed by pediatric ophthalmologist

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] FRAYSER R, HICKAM JB. EFFECT OF VASODILATOR DRUGS ON THE RETINAL BLOOD FLOW IN MAN. Arch Ophthalmol. 1965 May;73:640-2. doi: 10.1001/archopht.1965.00970030642008. No abstract available. PMID 14281979
- [Background] Yaster M, Simmons RS, Tolo VT, Pepple JM, Wetzel RC, Rogers MC. A comparison of nitroglycerin and nitroprusside for inducing hypotension in children: a double-blind study. Anesthesiology. 1986 Aug;65(2):175-9. doi: 10.1097/00000542-198608000-00008. PMID 3090906
- [Background] Dorner GT, Garhofer G, Kiss B, Polska E, Polak K, Riva CE, Schmetterer L. Nitric oxide regulates retinal vascular tone in humans. Am J Physiol Heart Circ Physiol. 2003 Aug;285(2):H631-6. doi: 10.1152/ajpheart.00111.2003. Epub 2003 May 15. PMID 12750062
- [Background] Munier FL, Beck-Popovic M, Balmer A, Gaillard MC, Bovey E, Binaghi S. Occurrence of sectoral choroidal occlusive vasculopathy and retinal arteriolar embolization after superselective ophthalmic artery chemotherapy for advanced intraocular retinoblastoma. Retina. 2011 Mar;31(3):566-73. doi: 10.1097/IAE.0b013e318203c101. PMID 21273941
- [Background] Shields CL, Bianciotto CG, Jabbour P, Ramasubramanian A, Lally SE, Griffin GC, Rosenwasser R, Shields JA. Intra-arterial chemotherapy for retinoblastoma: report No. 1, control of retinal tumors, subretinal seeds, and vitreous seeds. Arch Ophthalmol. 2011 Nov;129(11):1399-406. doi: 10.1001/archophthalmol.2011.150. Epub 2011 Jun 13. PMID 21670328
- [Background] Shields CL, Bianciotto CG, Jabbour P, Griffin GC, Ramasubramanian A, Rosenwasser R, Shields JA. Intra-arterial chemotherapy for retinoblastoma: report No. 2, treatment complications. Arch Ophthalmol. 2011 Nov;129(11):1407-15. doi: 10.1001/archophthalmol.2011.151. Epub 2011 Jun 13. PMID 21670326
- [Background] Fallaha N, Dubois J, Carret AS, Callejo SA, Hamel P, Superstein R. Real-time ophthalmoscopic findings of intraophthalmic artery chemotherapy in retinoblastoma. Arch Ophthalmol. 2012 Aug;130(8):1075-7. doi: 10.1001/archophthalmol.2012.180. No abstract available. PMID 22893086
- [Background] Cugati S, Varma DD, Chen CS, Lee AW. Treatment options for central retinal artery occlusion. Curr Treat Options Neurol. 2013 Feb;15(1):63-77. doi: 10.1007/s11940-012-0202-9. PMID 23070637
- [Background] Phillips TJ, McGuirk SP, Chahal HK, Kingston J, Robertson F, Brew S, Roebuck D, Hungerford JL, Herod J. Autonomic cardio-respiratory reflex reactions and superselective ophthalmic arterial chemotherapy for retinoblastoma. Paediatr Anaesth. 2013 Oct;23(10):940-5. doi: 10.1111/pan.12162. Epub 2013 May 13. PMID 23668238
- [Background] Kato MA, Green N, O'Connell K, Till SD, Kramer DJ, Al-Khelaifi M, Han JH, Pryor KO, Gobin YP, Proekt A. A retrospective analysis of severe intraoperative respiratory compliance changes during ophthalmic arterial chemosurgery for retinoblastoma. Paediatr Anaesth. 2015 Jun;25(6):595-602. doi: 10.1111/pan.12603. Epub 2015 Jan 7. PMID 25565164
- [Background] Scharoun JH, Han JH, Gobin YP. Anesthesia for Ophthalmic Artery Chemosurgery. Anesthesiology. 2017 Jan;126(1):165-172. doi: 10.1097/ALN.0000000000001381. No abstract available. PMID 27748655